CLINICAL TRIAL: NCT04207203
Title: Healthy Diet Rich in Potassium Containing Fruits, Vegetables and Nuts to Chronic Kidney Disease Patients Thought the Use of Sodium Zirconium Cyclosilicate: A Feasibility Study
Brief Title: Healthy Diet Rich in Potassium to Chronic Kidney Disease With Sodium Zirconium Cyclosilicate: A Feasibility Study
Acronym: HELPFUL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Peter Stenvinkel, Principal Investigator, Nephrologist, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ESR-18-13936
Record Dates: First submitted 2019-12-17; First posted 2019-12-20 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Chronic Kidney Disease stage4; Chronic Kidney Disease Stage 5; Hyperkalemia
Keywords: Healthy diet; Quality of life; Uremic toxins; Hyperkalemia; Chronic kidney disease; Gut microbiota
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperkalemia | interventions — sodium zirconium cyclosilicate; Diet, Healthy

STUDY DESIGN:
Intervention Model Description: In the first 3 weeks, stabilization phase, SZC will be prescribed to normalize plasma potassium to 3.5 to 5.0 mml/L, and a diet with energy 25-35 kcal/kg/day and protein 0.6 to 0.8 g/kg/day and with low K content will be prescribed. At the end of the first 3 weeks, the patients will initiate a healthy diet containing 3700 to 4000 mg/potassium for 3 weeks (healthy diet phase). A food basket containing fruits, vegetables, whole grains, nuts, white meat, fish and eggs in amounts adequate for the patient will be provided. Serum K will be monitored to promote serum K between 3.5 to 5.0 mmol/L and adjustments in the dose of SZC will be performed according to the drug label. During stabilization and healthy diet phases, serum K will be measured every 72 hours until serum K is normalized and after that, once per week.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm study (Other): During 3 weeks, SZC will be prescribed to normalize plasma potassium to 3.5 to 5.0 mml/L, and a diet with energy 25-35 kcal/kg/day and protein 0.6 to 0.8 g/kg/day and with low K content will be prescribed. At the end of the first 3 weeks, the patients will initiate a healthy diet containing 3700 to 4000 mg/potassium for 3 weeks (healthy diet phase). A food basket containing fruits, vegetables, whole grains, nuts, white meat, fish and eggs in amounts adequate for the patient will be provided. Serum K will be monitored to promote serum K between 3.5 to 5.0 mmol/L and adjustments in the dose of SZC will be performed according to the drug label. During stabilization and healthy diet phases, serum K will be measured every 72 hours until serum K is normalized and after that, once per week.
  Interventions: Combination Product: sodium zirconium cyclosilicate and healthy diet

INTERVENTIONS:
Combination Product: sodium zirconium cyclosilicate and healthy diet — During 3 weeks, SZC will be prescribed to normalize plasma potassium to 3.5 to 5.0 mml/L, and a diet with energy 25-35 kcal/kg/day and protein 0.6 to 0.8 g/kg/day and with low K content will be prescribed. At the end of the first 3 weeks, the patients will initiate a healthy diet containing 3700 to 4000 mg/potassium for 3 weeks (healthy diet phase). A food basket containing fruits, vegetables, whole grains, nuts, white meat, fish and eggs in amounts adequate for the patient will be provided. Serum K will be monitored to promote serum K between 3.5 to 5.0 mmol/L and adjustments in the dose of SZC will be performed according to the drug label. During stabilization and healthy diet phases, serum K will be measured every 72 hours until serum K is normalized and after that, once per week.

SUMMARY:
This is a descriptive single arm open-label interventional trial lasting 6 weeks aiming to test if a low protein healthy K-rich diet with fruits, vegetables, whole grains, and nuts with concomitant use of new potassium binder (SZC) can be safely prescribed to patients with chronic kidney disease (CKD) stages 4 and 5 with hyperkalemia. Thirty adult CKD patients with hyperkalemia will be included. In the first 3 weeks of the study the plasma K will be normalized with the use of SZC and then the participants will receive a fruit basket during 3 weeks. SZC will be continued thru out the study. Primary end points will be changes in patient satisfaction with treatment, patient symptom list, and intake of energy and protein before and after the stabilization and healthy diet phase. Secondary outcomes will include changes in quality of life, obstipation and circulating gut microbiota-related uremic toxins.

DETAILED DESCRIPTION:
Feasibility, descriptive single arm open-label interventional trial lasting 6 weeks. The study will recruit 36 CKD patients at the outpatient clinic with: age between 18 to 85 years; glomerular filtration rate < 29 ml/min/1.73 m2 and not on dialysis; serum K > 5.1 mmol/L or in previous use of sodium polystyrene sulfonate (SPS) to decrease serum K levels, and who develops hyperkalemia after SPS is ceased. Patients with serum K > 6.5 mmol/ and those likely to start dialysis within 2 months, with inflammatory bowel syndrome or with a history of hypokalemia (<3.0 mmol/L) will not be included. Primary end points will be changes in patient satisfaction with treatment, patient symptom list, and intake of energy and protein before and after the stabilization and healthy diet phase. Secondary outcomes will include changes in quality of life, obstipation and circulating gut microbiota-related uremic toxins. Intervention: In the first 3 weeks, representing stabilization phase, SZC will be prescribed to normalize plasma potassium to 3.5 to 5.0 mml/L, and a diet with energy 25-35 kcal/kg/day and protein 0.6 to 0.8 g/kg/day and with low K content will be prescribed by a renal dietitian. At the end of the first 3 weeks, the patients will be instructed to keep the diet with same content of energy and initiate a healthy diet containing 3700 to 4000 mg/potassium for 3 weeks (healthy diet phase). In order to increase adherence, a food basket containing fruits, vegetables, whole grains, nuts, white meat, fish and eggs in amounts adequate for the patient and the family will be provided. Serum K will be monitored to promote serum K between 3.5 to 5.0 mmol/L and adjustments in the dose of SZC will be performed according to the drug label. Blood measurements, questionnaires related to quality of life and intestinal obstipation and measurements of nutritional intake will be performed in the beginning and at the end of the stabilization phase and again in the beginning and end of the healthy diet phase. Additionally, during stabilization and healthy diet phases, serum K will be measured every 72 hours until serum K is normalized and after that, once per week.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 to 85 years; glomerular filtration rate < 29 ml/min/1.73 m2 and not on dialysis; serum K > 5.1 mmol/L or in previous use of sodium polystyrene sulfonate (SPS) to decrease serum K levels, and who develops hyperkalemia after SPS is ceased.

Exclusion Criteria:

* Patients with serum K > 6.5 mmol/ and those likely to start dialysis within 2 months, with inflammatory bowel syndrome or with a history of hypokalemia (<3.0 mmol/L). Pregnant women.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-11-03 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-05-10 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction | 6 weeks
  Renal Treatment Satisfaction Questionnaire (RTSQ). It si based on 13 questions, each varying from 0 to 6. Total score is 78, being the highest score the better.
Symptoms list | 6 weeks
  Symptoms list
Energy intake | 6 weeks
  24-hour food recalls
Protein intake | 6 weeks
  24-hour food recalls

SECONDARY OUTCOMES:
Plasma potassium | 6 weeks
  Plasma potassium concentration
Short Form Health Survey (SF-36) | 6 weeks
  Short Form Health Survey (SF-36). It is calculated using norm-based scoring, which employs linear transformation to achieve standardized scores with a mean of 50. the highest, the better.
Intestinal obstipation | 6 weeks
  Bristol stool chart
Inflammatory marker 1 | 6 weeks
  C-reactive protein concentration
Inflammatory marker 2 | 6 weeks
  Interleukin 6 concentration
Microbiota-derived uremic retention solutes 1 | 6 weeks
  P-cresyl sulfate concentration
Microbiota-derived uremic retention solutes 2 | 6 weeks
  Indoxyl-sulfate concentration
Microbiota-derived uremic retention solutes 3 | 6 weeks
  Trimethylamine N-oxide concentration

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers

REFERENCES:
- [Derived] Avesani CM, Heimburger O, Rubin C, Sallstrom T, Faxen-Irving G, Lindholm B, Stenvinkel P. Plant-based diet in hyperkalemic chronic kidney disease patients receiving sodium zirconium cyclosilicate: a feasibility clinical trial. Am J Clin Nutr. 2024 Sep;120(3):719-726. doi: 10.1016/j.ajcnut.2024.06.025. Epub 2024 Jul 18. PMID 39032787